CLINICAL TRIAL: NCT02396992
Title: Evaluation of a Minimal-massive Intervention in Elderly Hospitalized Patients With Oropharyngeal Dysphagia
Brief Title: Minimal-Massive Intervention in Elderly Patients With Dysphagia
Acronym: MMI
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hospital de Mataró (Other)
Responsible Party: Principal Investigator, Pere Clave, PhD. MD surgery., Hospital de Mataró
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: IMM2013-14
Record Dates: First submitted 2014-06-25; First posted 2015-03-24 (Estimated); Last update posted 2019-05-01 (Actual); Status verified 2019-04

CONDITIONS: Oropharyngeal Dysphagia
Keywords: Oropharyngeal Dysphagia; Aspiration pneumonia; Malnutrition; Oral Health; Bacterial colonization; Aging
MeSH Terms: conditions — Deglutition Disorders; Pneumonia, Aspiration; Malnutrition

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Minimal-Massive Intervention (Other): The minimal/basic intervention for a massive number of hospitalized patients.
  Interventions: Other: Minimal-Massive Intervention

INTERVENTIONS:
Other: Minimal-Massive Intervention — The intervention will consist in basic recommendations based on the evaluations done at admission and discharge: a) diet adaptation (solids and fluids) based on dysphagia clinical evaluation (V-VST) to avoid efficacy or safety alterations; b) nutritional supplements in case of malnutrition (MNA-sf; bioimpedance and blood analysis) to improve nutritional status;and c) oral health and hygiene recommendations (toothbrushing and antiseptic mouthwashes to decline bacterial colonization).

SUMMARY:
The purpose of this study is to apply a minimal-massive intervention (minimal recommendations to maximal number of patients) to elderly (>70 years) hospitalized patients with oropharyngeal dysphagia (OD). The intervention will consist of early screening and assessment of OD, malnutrition and oral hygiene. Patients will be given recommendations for adaptation of volume and viscosity of fluids, nutritional support and good oral hygiene practices and followed at 3, 6, 9 and 12 months after discharge. In every point of the follow-up period, patients will be re-evaluated to adjust recommendations and to verify their compliance with the treatment.

The objectives of the intervention are to have an impact on complications related to OD (avoid impaired safety alterations and improve nutritional and oral health status and reduce) and to reduce readmissions, readmissions for pneumonia and morbimortality.

DETAILED DESCRIPTION:
These study aims to evaluate the application of an assistance programme to:

1. Perform a systematic screening of oropharyngeal dysphagia in older hospitalized patients (≥70 yr) admitted to internal medicine and geriatric unit of Hospital de Mataró.
2. Offer a minimal-massive treatment to older patients with OD based on, rheological adaptation of fluids (volume and viscosity), nutritional support based on traditional diet and oral hygiene treatment.
3. To give education and knowledge about the diagnose and treatment of OD to the medical staff, caregivers and relatives of the patients to improve their management.

Study design:

Experimental pre-post interventional study with 1 year follow-up and 4 control points at 3, 6, 9 and 12 months after discharge. Pre-interventional evaluations will be done on admission and at discharge; post-interventional evaluations will be performed at 3, 6, 9 and 12 months after discharge. In every evaluation point the investigators will obtain data about OD (efficacy and safety of swallow with the Volume-Viscosity Swallowing Test (V-VST)), health status of the patients (comorbidities, functionality, frailty, anthropometric measurements, illnesses and medication), nutritional status (MNA-sf and Bioimpedance), oral hygiene (dental evaluation with the Simplified Oral Hygiene Index (OHI-S)) and respiratory infections and pneumonia rates. In addition during the follow-up period the investigators will collect readmissions incidence (all readmissions, respiratory infections and pneumonia), institutionalization and death. Data collected will be compared with the previous year of the same patient and with a historical control group of untreated older patients with OD that will be matched for age, sex, comorbidities and functionality.

The intervention will consist on adaptation of fluids (volume and viscosity) in accordance with V-VST results, nutritional supplementation with traditional food (based on MNA-sf and bioimpedance results) and recommendation of good oral hygiene practices (based on dental evaluation). In every point of the follow-up period, recommendations will be given to patients.

Objectives:

* The primary objective is to launch and evaluate the effect of the minimal-massive program in hospitalized older patients with OD.
* To evaluate the effect of the intervention on the signs and symptoms of OD, nutritional status, oral hygiene, functional status and quality of life of patients included at the program at 3, 6, 9 and 12 months after discharge.
* To describe readmission rates for any reason, readmission rates for pneumonia, institutionalization rate and mortality rate in the study population compared to an historical control group of older patients with OD and no intervention.

ELIGIBILITY:
Inclusion Criteria:

* Older patients (≥70 years) admitted to Unit 5 and 8 of Hospital de Mataró.
* With OD diagnosed by the V-VST.
* Patients that have signed the informed consent form.
* Patients without any exclusion criteria.

Exclusion Criteria:

* Patients not able to comply with the protocol.
* Patients currently participating in any clinical trial or during the 4 last weeks.
* Patients with severe dementia or inability to communicate (GDS ≥ 6).
* Patients of the Intensive Care Unit.
* Patients with low functionality (Barthel pre-admission ≤ 40).
* Patients with high mortality risk (Walter score > 6).

Min Age: 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 62 (Actual)
Dates: Start 2014-03; Primary Completion 2015-06 (Actual); Study Completion 2015-09 (Actual)

PRIMARY OUTCOMES:
Reduction of incidence of respiratory infections due to the intervention. | One year after discharge
  Readmissions for respiratory infections (including pneumonia) will be recorded and compared with the previous year of the same patient (pre-post study) and with a retrospective control group of elderly patients with dysphagia without intervention. Review of the medical history of the patient will be done by a medical doctor. Follow-up visits will be done every three months for a total of 12 months.

SECONDARY OUTCOMES:
Improvement of signs and symptoms of oropharyngeal dysphagia | One year after discharge
  To evaluate the effects of the minimal-massive intervention above signs and symptoms of oropharyngeal dysphagia due to the use of thickener. Follow-up visits will be done every three months for a total of 12 months.
Improvement of nutritional status of the patients enrolled. | One year after discharge
  To evaluate the effects of the minimal-massive intervention above nutritional status of the patient measured with the MNA-sf, bioimpedance and blood analytical parameters. Follow-up visits will be done every three months for a total of 12 months.
Improvement of oral health and hygiene of the patients enrolled. | One year after discharge
  To evaluate the effects of the minimal-massive intervention above oral hygiene status of the patients measured with the OHI-S and a dental examination including periodontal disease and caries. Follow-up visits will be done every three months for a total of 12 months.
Improvement of quality of life of patients enrolled. | One year after discharge
  To evaluate the effects of the minimal-massive intervention in quality of life of patients enrolled measured with the EQ5D questionnaire.

CONTACTS AND LOCATIONS:
Overall Officials: Pere Clavé, PhD; MD, Principal Investigator — Hospital de Mataró
Locations (1):
- Hospital de Mataró. Consorci Sanitari del Maresme., Mataró, Barcelona, Spain

REFERENCES:
- [Derived] Martin A, Ortega O, Roca M, Arus M, Clave P. Effect of A Minimal-Massive Intervention in Hospitalized Older Patients with Oropharyngeal Dysphagia: A Proof of Concept Study. J Nutr Health Aging. 2018;22(6):739-747. doi: 10.1007/s12603-018-1043-3. PMID 29806864